CLINICAL TRIAL: NCT05523934
Title: Capsaïcin patch8% in Adult Complex Regional Pain Syndromes: a Retrospective Analysis
Brief Title: Retrospective Analysis of capsaïcin Patch in Complex Regional Pain Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of department, anesthesiology, Brugmann University Hospital
Other Study IDs: patch_CRPS-retro
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Capsaïcine patch — Patients with complex regional pain syndrome under maximal conventional treatment having a supplementary treatment by a capsaïcin patch.

SUMMARY:
Complex regional pain syndrome is a painful syndrome often secondary to a traumatic lesion. Treatment is difficult, of long duration with variable outcomes. Patch of capsaïcin has been proposed as adjuvant to a multimodal treatment. Capsaïcin may act by its effect on transient receptor potential vanilloid 1. Efficacity and outcome studies with this treatment are lacking.

The aim of this retrospective study is to evaluate pain intensity over time assessed by visual analog scale in patient with complex regional pain syndrome treated with capsaïcin patch in addition to their usual treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with complex regional pain syndrome on maximum medical treatment
* Age ≥18 years
* Patients treated between 2012 and August 31, 2022 in the pain clinic of the CHU Brugmann

Exclusion Criteria:

- incomplete medical chart

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients treated between 2012 and 2022 in the Pain Clinic of the CHU Brugmann for complex regional pain syndrome and who have been treated by a capsaïcin patch in addition to their normal treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 month period
  Pain intensity evaluated by a visual analog scale (on a scale 0 to 10) by patients before and after capsaïcin addition.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Besse, MD, Study Chair — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baron R, Fields HL, Janig W, Kitt C, Levine JD. National Institutes of Health Workshop: reflex sympathetic dystrophy/complex regional pain syndromes--state-of-the-science. Anesth Analg. 2002 Dec;95(6):1812-6. doi: 10.1097/00000539-200212000-00064. No abstract available. PMID 12456464
- [Background] Birklein F. Complex regional pain syndrome. J Neurol. 2005 Feb;252(2):131-8. doi: 10.1007/s00415-005-0737-8. PMID 15729516
- [Background] Geertzen JH, Dijkstra PU, Groothoff JW, ten Duis HJ, Eisma WH. Reflex sympathetic dystrophy of the upper extremity--a 5.5-year follow-up. Part I. Impairments and perceived disability. Acta Orthop Scand Suppl. 1998 Apr;279:12-8. PMID 9614810
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Steyaert A, Lavand'homme P. Prevention and Treatment of Chronic Postsurgical Pain: A Narrative Review. Drugs. 2018 Mar;78(3):339-354. doi: 10.1007/s40265-018-0866-x. PMID 29380289
- [Background] Arora V, Campbell JN, Chung MK. Fight fire with fire: Neurobiology of capsaicin-induced analgesia for chronic pain. Pharmacol Ther. 2021 Apr;220:107743. doi: 10.1016/j.pharmthera.2020.107743. Epub 2020 Nov 10. PMID 33181192
- [Background] Simpson DM, Robinson-Papp J, Van J, Stoker M, Jacobs H, Snijder RJ, Schregardus DS, Long SK, Lambourg B, Katz N. Capsaicin 8% Patch in Painful Diabetic Peripheral Neuropathy: A Randomized, Double-Blind, Placebo-Controlled Study. J Pain. 2017 Jan;18(1):42-53. doi: 10.1016/j.jpain.2016.09.008. Epub 2016 Oct 13. PMID 27746370
- [Background] Backonja M, Wallace MS, Blonsky ER, Cutler BJ, Malan P Jr, Rauck R, Tobias J; NGX-4010 C116 Study Group. NGX-4010, a high-concentration capsaicin patch, for the treatment of postherpetic neuralgia: a randomised, double-blind study. Lancet Neurol. 2008 Dec;7(12):1106-12. doi: 10.1016/S1474-4422(08)70228-X. Epub 2008 Oct 30. PMID 18977178
- [Background] Simpson DM, Brown S, Tobias J; NGX-4010 C107 Study Group. Controlled trial of high-concentration capsaicin patch for treatment of painful HIV neuropathy. Neurology. 2008 Jun 10;70(24):2305-13. doi: 10.1212/01.wnl.0000314647.35825.9c. PMID 18541884
- [Background] Babbar S, Marier JF, Mouksassi MS, Beliveau M, Vanhove GF, Chanda S, Bley K. Pharmacokinetic analysis of capsaicin after topical administration of a high-concentration capsaicin patch to patients with peripheral neuropathic pain. Ther Drug Monit. 2009 Aug;31(4):502-10. doi: 10.1097/FTD.0b013e3181a8b200. PMID 19494795
- [Background] Simpson DM, Gazda S, Brown S, Webster LR, Lu SP, Tobias JK, Vanhove GF; NGX-4010 C118 Study Group. Long-term safety of NGX-4010, a high-concentration capsaicin patch, in patients with peripheral neuropathic pain. J Pain Symptom Manage. 2010 Jun;39(6):1053-64. doi: 10.1016/j.jpainsymman.2009.11.316. PMID 20538187
- [Background] Frias B, Merighi A. Capsaicin, Nociception and Pain. Molecules. 2016 Jun 18;21(6):797. doi: 10.3390/molecules21060797. PMID 27322240
- [Background] Basith S, Cui M, Hong S, Choi S. Harnessing the Therapeutic Potential of Capsaicin and Its Analogues in Pain and Other Diseases. Molecules. 2016 Jul 23;21(8):966. doi: 10.3390/molecules21080966. PMID 27455231
- [Background] Caterina MJ, Leffler A, Malmberg AB, Martin WJ, Trafton J, Petersen-Zeitz KR, Koltzenburg M, Basbaum AI, Julius D. Impaired nociception and pain sensation in mice lacking the capsaicin receptor. Science. 2000 Apr 14;288(5464):306-13. doi: 10.1126/science.288.5464.306. PMID 10764638
- [Background] Chen W, Chi YN, Kang XJ, Liu QY, Zhang HL, Li ZH, Zhao ZF, Yang Y, Su L, Cai J, Liao FF, Yi M, Wan Y, Liu FY. Accumulation of Cav3.2 T-type Calcium Channels in the Uninjured Sural Nerve Contributes to Neuropathic Pain in Rats with Spared Nerve Injury. Front Mol Neurosci. 2018 Feb 8;11:24. doi: 10.3389/fnmol.2018.00024. eCollection 2018. PMID 29472842
- [Background] Jancso G, Santha P. The foundation of sensory pharmacology: Nicholas (Miklos) Jancso and the Szeged contribution. Temperature (Austin). 2015 May 26;2(2):152-7. doi: 10.1080/23328940.2015.1045683. eCollection 2015 Apr-Jun. PMID 27227015
- [Background] Chung MK, Campbell JN. Use of Capsaicin to Treat Pain: Mechanistic and Therapeutic Considerations. Pharmaceuticals (Basel). 2016 Nov 1;9(4):66. doi: 10.3390/ph9040066. PMID 27809268